CLINICAL TRIAL: NCT01507116
Title: Diabetes Attitudes Wishes and Needs (DAWN) 2 Study: A Multinational, Multi-stakeholder Survey Study of Psychosocial Issues in Diabetes and Patient-centred Diabetes Care
Brief Title: Diabetes Attitudes Wishes and Needs
Acronym: DAWN2
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3966; U1111-1123-7509 (Other: WHO)
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Relatives to/Carers of Patients; Healthcare Professionals
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- People with Diabetes
  Interventions: Other: No treatment given
- Family Members
  Interventions: Other: No treatment given
- Healthcare Professionals
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Three separate survey questionnaires, one for each of the three diabetes groups. Each questionnaire is composed of multiple items including pre-coded (multiple choice) questions, dichotomous (yes/no) questions and rating scales.

SUMMARY:
The study is conducted in Africa, Asia, Europe, Japan, North America and South America.

The multinational surveys will explore the experiences and unmet needs of people with diabetes, as well as those of family members of people with diabetes, and of healthcare professionals treating people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 18 years with diabetes (type 1 or type 2: not only during pregnancy)
* Adults aged at least 18 years involved in the daily care of an adult (18 years or older) with diabetes (type 1 or type 2)
* General practitioners who personally treat at least 5 adults (18 years or older) with diabetes per month and initiate oral medication
* Diabetes specialists (endocrinologists/diabetologists) who personally treat at least 50 adults (18 years or older) with diabetes per month and prescribe oral medication, insulin or other injectable diabetes medications
* Diabetes educators (diabetes nurses/dieticians/other non-physician healthcare professionals) providing care for at least 5 adults (18 years or older) with diabetes per month
* Participants must have access to the internet, either at home or at a location convenient to them, or be able to attend a face-to-face or telephone interview, to participate in the survey
* Provision of informed consent before the start of any study-related activities

Exclusion Criteria:

* Individuals aged below 18 years and/or diagnosed with diabetes less than 12 months ago
* Inability to understand and comply with written and verbal instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total core study population is intended to comprise 9540 people with diabetes, 2160 family members and 5040 healthcare professionals across the 18 countries participating in DAWN 2. The study population will be invited to participate by either web based or telephone recruitment, or if absolutely needed and deemed appropriate, physician recruitment (i.e. patients recruited by physicians will telephone call centres managed by the local survey research agency and will be screened by telephone).
Sampling Method: Non-Probability Sample
Enrollment: 8985 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Self-reported health and Quality of Life (QoL) (measured by the study questionnaire) | Day 1

SECONDARY OUTCOMES:
Psychological well-being of people with diabetes and family members measured by the study questionnaire | Day 1
Diabetes distress of people with diabetes and family members measured by the study questionnaire | Day 1
Self-reported self-management of people with diabetes measured by the study questionnaire | Day 1
Family support behaviours reported by people with diabetes and family members measured by the study questionnaire | Day 1
Patient-centred diabetes care reported by people with diabetes and health care professionals measured by the study questionnaire | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Algiers, Algeria
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China
- Novo Nordisk Investigational Site, Copenhagen S, Denmark
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Tokyo, Japan
- Novo Nordisk Investigational Site, Mexico City, Mexico
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Peyrot M, Burns KK, Davies M, Forbes A, Hermanns N, Holt R, Kalra S, Nicolucci A, Pouwer F, Wens J, Willaing I, Skovlund SE. Diabetes Attitudes Wishes and Needs 2 (DAWN2): a multinational, multi-stakeholder study of psychosocial issues in diabetes and person-centred diabetes care. Diabetes Res Clin Pract. 2013 Feb;99(2):174-84. doi: 10.1016/j.diabres.2012.11.016. Epub 2012 Dec 27. PMID 23273515
- [Result] Nicolucci A, Kovacs Burns K, Holt RI, Comaschi M, Hermanns N, Ishii H, Kokoszka A, Pouwer F, Skovlund SE, Stuckey H, Tarkun I, Vallis M, Wens J, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national benchmarking of diabetes-related psychosocial outcomes for people with diabetes. Diabet Med. 2013 Jul;30(7):767-77. doi: 10.1111/dme.12245. PMID 23711019
- [Result] Kovacs Burns K, Nicolucci A, Holt RI, Willaing I, Hermanns N, Kalra S, Wens J, Pouwer F, Skovlund SE, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national benchmarking indicators for family members living with people with diabetes. Diabet Med. 2013 Jul;30(7):778-88. doi: 10.1111/dme.12239. PMID 23701236
- [Result] Holt RI, Nicolucci A, Kovacs Burns K, Escalante M, Forbes A, Hermanns N, Kalra S, Massi-Benedetti M, Mayorov A, Menendez-Torre E, Munro N, Skovlund SE, Tarkun I, Wens J, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national comparisons on barriers and resources for optimal care--healthcare professional perspective. Diabet Med. 2013 Jul;30(7):789-98. doi: 10.1111/dme.12242. PMID 23710839
- [Result] Funnell M. Beyond the data: moving towards a new DAWN in diabetes. Diabet Med. 2013 Jul;30(7):765-6. doi: 10.1111/dme.12244. No abstract available. PMID 23710971
- [Result] Peyrot M, Egede LE, Campos C, Cannon AJ, Funnell MM, Hsu WC, Ruggiero L, Siminerio LM, Stuckey HL. Ethnic differences in psychological outcomes among people with diabetes: USA results from the second Diabetes Attitudes, Wishes, and Needs (DAWN2) study. Curr Med Res Opin. 2014 Nov;30(11):2241-54. doi: 10.1185/03007995.2014.947023. Epub 2014 Aug 18. PMID 25079662
- [Derived] Peyrot M, Egede LE, Funnell MM, Hsu WC, Ruggiero L, Siminerio LM, Stuckey HL. US ethnic group differences in self-management in the 2nd diabetes attitudes, wishes and needs (DAWN2) study. J Diabetes Complications. 2018 Jun;32(6):586-592. doi: 10.1016/j.jdiacomp.2018.03.002. Epub 2018 Mar 8. PMID 29709335
- [Derived] Nefs G, Pouwer F. The role of hypoglycemia in the burden of living with diabetes among adults with diabetes and family members: results from the DAWN2 study in The Netherlands. BMC Public Health. 2018 Jan 18;18(1):156. doi: 10.1186/s12889-018-5064-y. PMID 29347915
- [Derived] Barnard KD, Holt RI, Dyson PA, Cummings MH, Kanumilli N, O'Neill S, Hall G. Could the Discrepancy in Perceived Emotional Care Received and Provided Be a Barrier to Active Diabetes Self-management? Insights From the Second Diabetes Attitudes, Wishes and Needs (DAWN2) Study. Diabetes Care. 2016 Feb;39(2):e20-1. doi: 10.2337/dc15-0674. Epub 2015 Dec 30. No abstract available. PMID 26721814
- [Derived] Peyrot M, Egede LE, Funnell MM, Hsu WC, Ruggiero L, Siminerio LM, Stuckey HL. Ethnic differences in family member diabetes involvement and psychological outcomes: results from the second Diabetes Attitudes, Wishes and Needs (DAWN2) study in the USA. Curr Med Res Opin. 2015;31(7):1297-307. doi: 10.1185/03007995.2015.1043251. Epub 2015 May 20. PMID 25907127
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com